CLINICAL TRIAL: NCT05762172
Title: Interest of the Early Dynamic F-DOPA PET Examination for Differential Diagnosis Between Recurrence and Radionecrosis of Brain Metastasis
Brief Title: Dynamic F-DOPA PET for Differential Diagnosis Between Recurrence and Radionecrosis of Brain Metastasis
Acronym: DYNDOPATEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2022_843_0055
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Brain Metastases; Radiation Necrosis
Keywords: silicon PET/CT; 18F-DOPA; short time examination; Brain Metastases; Radiation Necrosis
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: early 18F-FDOPA uptake — During the usual patient care protocol for the 18F-FDOPA TEP examination, a 10 min acquisition starts after a 15 minutes waiting period following the injection of the radiotracer. This allows the reconstruction of a single late image volume. In the framework of this project, the patient is placed in the machine at the time of injection so as to acquire early 18F-FDOPA uptake and then reconstruct intermediate image volumes in addition to the usual final volume.
  The total duration of the patient's examination is therefore not changed.

SUMMARY:
Contrast-enhanced magnetic resonance imaging is the most widely used examination for detecting the presence of brain metastasis. Functional sequences such as perfusion weighted imaging makes it possible to differentiate tumor recurrence from cerebral radionecrosis. However, this imaging technique may exhibit limitations, especially for brain lesions consisting of a mixture of necrotic tissue and tumor progression or depending on the location of the lesion in the brain. The use of 18F-DOPA PET is another option available to oncologists. Many studies on gliomas showed the superiority of this imaging technique over contrast-enhanced MRI. However, this imaging solution has been very poorly studied for brain metastases. The new PET technology equiped with silicon detectors makes it possible to obtain greater sensitivities than those of previous generations. It also make possible to obtain images in very short acquisition times. After injection, the hardware allows to obtain the perfusion kinetics of the lesion thanks to a very short temporal sampling (i.e. three seconds).

The main objective of this pilot study is to evaluate the association between early activity measurements (< 4 minutes post-injection) of 18F-FDOPA in PET and the differential diagnosis between radionecrosis and recurrence of cerebral metastases treated by radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for cerebral 18F-FDOPA PET examination prescribed as part of his usual medical care for brain metastasis
* Age ≥ 18 years old
* Affiliation to a social security program
* Ability of the subject to understand and express opposition

Exclusion Criteria:

* Age under 18
* Person under guardianship or curators
* Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
difference between the maximum activity (in Bq/mL) in the venous sinus and the maximum activity present in the region of interest encompassing the lesion being studied. | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bailly P, Bouzerar R, Barrat I, Boone M, Coutte A, Meyer ME. A Practical, Short, [18F]F-DOPA PET/CT Acquisition Method for Distinguishing Recurrent Brain Metastases from Radionecrosis Following Radiotherapy. J Clin Med. 2025 Mar 22;14(7):2168. doi: 10.3390/jcm14072168. PMID 40217619